CLINICAL TRIAL: NCT00003855
Title: A Randomized Trial of Axillary Node Dissection in Women With Clinical T1-2 N0-1 M0 Breast Cancer Who Have a Positive Sentinel Node
Brief Title: Lymph Node Removal in Treating Women Who Have Stage I or Stage IIA Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACOSOG-Z0011; GUMC-00153; CDR0000067018 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Breast Cancer
Keywords: stage IA breast cancer; stage IB breast cancer; stage II breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgery + radiotherapy (Experimental): Patients undergo axillary lymph node dissection involving removal of at least level I and II nodes, followed by whole-breast radiotherapy (exclusive of a third supraclavicular field) 5 days a week for a maximum of 7 weeks. Patients may receive adjuvant systemic therapy at the discretion of the treating physician.
  Patients are followed up at 30 days, at 6, 12, 18, 30, and 36 months, and then annually for a total of 10 years.
  Interventions: Procedure: axillary lymph node dissection; Radiation: whole breast irradiation
- Radiotherapy (Active Comparator): Patients undergo breast radiotherapy only. Patients may receive adjuvant systemic therapy at the discretion of the treating physician.
  Patients are followed up at 30 days, at 6, 12, 18, 30, and 36 months, and then annually for a total of 10 years.
  Interventions: Radiation: whole breast irradiation

INTERVENTIONS:
Procedure: axillary lymph node dissection
  Arms: Surgery + radiotherapy
Radiation: whole breast irradiation

SUMMARY:
RATIONALE: Surgery to remove lymph nodes in the armpit may remove cancer cells that have spread from tumors in the breast.

PURPOSE: Randomized phase III trial to determine the effectiveness of removing lymph nodes in the armpit in treating women who have stage I or stage IIA breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary objectives:

Long term: To assess whether overall survival for patients randomized to Arm 2 (no immediate ALND) is essentially equivalent to (or better than) than that for patients assigned to Arm 1 (completion ALND).

Short term: To quantify and compare the surgical morbidities associated with SLND plus ALND versus SLND alone.

OUTLINE: This is a randomized study. After segmental mastectomy and sentinel lymph node dissection, patients are stratified according to age (50 and under vs over 50), estrogen receptor status (positive vs negative), and tumor size (no greater than 1 cm vs greater than 1 cm but no greater than 2 cm vs greater than 2 cm). Patients are randomized to one of two treatment arms.

ELIGIBILITY:
Inclusion Criteria:

PLEASE NOTE: Patients registered to this study may undergo intra-operative or post¬operative randomization.

1. Patient must be female.
2. Patient must be at least 18 years of age.
3. Patient's clinical stage must be documented as tumor size less than 5 cm, with no palpable nodes and no evidence of metastatic disease (T1 or T2 N0 M0; see appendices for staging criteria) and the tumor documented as amenable to lumpectomy.
4. Patient must have a tissue diagnosis of invasive breast carcinoma. Note: A patient can be registered to this study if they have a cytologic diagnosis suggestive of carcinoma from a fine needle aspiration (FNA) of a palpable or non-palpable breast lesion and the investigator believes the breast lesion is clinically suspicious for invasive breast carcinoma.
5. Date of the patient's first tissue diagnosis of invasive breast carcinoma or cytologic diagnosis of carcinoma must be no more than 60 days prior to the SLND.
6. The patient who had BCT (segmental mastectomy) performed previously, and is now referred to the local investigator for SLND, is eligible if the BCT was less than or equal to 60 days prior to the SLND. NOTE: Copies of the operative and pathology reports must be submitted as part of the registration process.
7. Patient must have ECOG/Zubrod status =2, as documented in patient's medical record.
8. Patient must be available for follow-up.
9. Patient of childbearing potential must have a negative serum or urine pregnancy test within 14 days of beginning study interventions.
10. Patient must have access to radiation therapy.
11. A sentinel lymph node must be identified that contains metastatic breast cancer as documented by frozen section, touch prep, or H&E staining on permanent section.

    * NOTE: Patients with metastatic breast cancer identified by immunohistochemistry (IHC) are not eligible.
12. Patient randomized to ALND must undergo ALND within 42 days of their SLND.
13. A patient with a history of a previous malignancy is eligible for this study as long as the patient meets the following criteria for a cancer survivor. A cancer survivor is eligible provided that the following criteria are met:

    1. The patient has undergone potentially curative therapy for all prior malignancies,
    2. There has been no evidence of any prior malignancies for at least five years with no evidence of recurrence (except for effectively treated basal cell or squamous carcinoma of the skin, carcinoma in -situ of the cervix that has been effectively treated by surgery alone, or lobular carcinoma in-situ of the ipsilateral or contralateral breast treated by surgery alone), and
    3. The patient is deemed by their treating physician to be at low risk for recurrence from prior malignancies.
14. Patient or the patient's legally acceptable representative must provide a signed and dated written informed consent prior to registration and any study-related procedures.
15. Patient must provide written authorization to allow the use and disclosure of their protected health information. NOTE: This may be obtained in either the study-specific informed consent or in a separate authorization form and must be obtained from the patient prior to study registration.

Exclusion Criteria:

1. Patient is lactating (breastfeeding).
2. Patient has been previously treated with chemotherapy, estrogen receptor antagonists (i.e., Tamoxifen) or selective estrogen receptor modulators (SERMs, i.e., Raloxifene) for this invasive breast cancer.
3. Patient has a previously placed pre-pectoral breast implant. NOTE: A subpectoral implant is allowed.
4. Patient has concurrent invasive bilateral breast malignancies.
5. Patient has clinically and radiologically identified multi-centric disease that is not amenable to a single lumpectomy.
6. Patient has had previous ipsilateral axillary surgery such as excisional biopsy of lymph node(s), treatment of hidradenitis.
7. Patient has a medical contraindication to ALND or is considered a poor surgical risk due to a non-malignant systemic disease (cardiovascular, renal, etc.) that would preclude the treatment options.
8. Patient who is noted to have matted nodes or gross extranodal disease at the time of SLND.
9. Patient has three or more positive sentinel nodes by frozen section, touch prep, or H&E staining on permanent section.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 605 (Actual)
Dates: Start 1999-04; Primary Completion 2007-08 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Overall survival | Up to 10 years
Morbidity | Up to 10 years
Disease-free survival | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Armando E. Giuliano, MD, Study Chair — Saint John's Cancer Institute
Locations (156):
- United States (152):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Providence Cancer Center, Mobile, Alabama
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - CCOP - Mayo Clinic Scottsdale Oncology Program, Scottsdale, Arizona
  - Washington Regional Medical Center, Fayetteville, Arkansas
  - St. Vincent Doctors Doctors Hospital, Little Rock, Arkansas
  - Baptist Health Medical Center, Little Rock, Arkansas
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Mercy San Juan Hospital, Carmichael, California
  - Arrowhead Regional Medical Center, Colton, California
  - Mount Diablo Regional Cancer Center, Concord, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Summit Medical Center, Oakland, California
  - St. Joseph Hospital Regional Cancer Center - Orange, Orange, California
  - Palo Alto Medical Foundation, Palo Alto, California
  - Huntington Cancer Center at Huntington Hospital, Pasadena, California
  - Shasta Regional Medical Center, Redding, California
  - University of California Davis Cancer Center, Sacramento, California
  - Sharp Memorial Hospital, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - John Wayne Cancer Institute at Saint John's Health Center, Santa Monica, California
  - Sonoma Valley Hospital, Sonoma, California
  - St. Joseph's Regional Cancer Center, Stockton, California
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Aurora, Colorado
  - Memorial Hospital Cancer Center, Colorado Springs, Colorado
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Morton Plant Hospital, Clearwater, Florida
  - Lakeland Regional Cancer Center at Lakeland Regional Medical Center, Lakeland, Florida
  - Watson Clinic, Lakeland, Florida
  - Martin Memorial Cancer Center, Stuart, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Albany, Georgia
  - Phoebe Cancer Center at Phoebe Putney Memorial Hospital, Albany, Georgia
  - Charles B. Eberhart Cancer Center at DeKalb Medical Center, Decatur, Georgia
  - Surgical Oncology of Northeast Georgia, Gainesville, Georgia
  - St. Francis Medical Center, Honolulu, Hawaii
  - Kaiser Permanente Medical Center, Honolulu, Hawaii
  - St. Luke's Regional Medical Center, Boise, Idaho
  - St. Elizabeth's Hospital, Belleville, Illinois
  - Belleville Memorial Hospital, Belleville, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois
  - Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - Evanston Northwestern Health Care - Evanston Hospital, Evanston, Illinois
  - St. Francis Hospital and Health Centers, Beech Grove, Indiana
  - Deaconess Hospital, Evansville, Indiana
  - St. Mary's Medical Center, Evansville, Indiana
  - Central Baptist Hospital, Lexington, Kentucky
  - Norton Healthcare Cancer Center, Louisville, Kentucky
  - Woman's Hospital, Baton Rouge, Louisiana
  - Baton Rouge General Regional Cancer Center, Baton Rouge, Louisiana
  - Maine Medical Center, Portland, Maine
  - DeCesaris Cancer Institute at Anne Arundel Medical Center, Annapolis, Maryland
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Fallon Clinic at Worcester Medical Center, Worcester, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Health System, Detroit, Michigan
  - Great Lakes Cancer Institute - McLaren, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Butterworth Hospital, Grand Rapids, Michigan
  - Spectrum Health Downtown Campus, Grand Rapids, Michigan
  - Spectrum Health - Blodgett Campus, Grand Rapids, Michigan
  - Henry Ford Medical Center - West Bloomfield, West Bloomfield, Michigan
  - Park Nicollet Clinic, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Keesler Medical Center - Keesler Air Force Base, Keesler Air Force Base, Mississippi
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - St. Louis University Hospital Cancer Center, St Louis, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Southern New Hampshire Medical Center, Nashua, New Hampshire
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital, Marlton, New Jersey
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Lutheran Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Louis Busch Hager Cancer Center at Mary Imogene Bassett Hospital, Cooperstown, New York
  - Kingston Hospital, Kingston, New York
  - Fern Feldman Anolick Breast Center at Benedictine Hospital, Kingston, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Highland Hospital of Rochester, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Comprehensive Cancer Center at Our Lady of Mercy Medical Center, The Bronx, New York
  - Hope A Women's Cancer Center, Asheville, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Tri-Health Good Samaritan Hospital, Cincinnati, Ohio
  - Ireland Cancer Center at University Hospitals of Cleveland and Case Western Reserve University, Cleveland, Ohio
  - Arthur G. James Cancer Hospital at Ohio State University, Columbus, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - Flower Hospital - ProMedica Health System, Sylvania, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Kaiser Permanente Medical Office - Mother Joseph Plaza, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Sacred Heart Hospital, Allentown, Pennsylvania
  - John and Dorothy Morgan Cancer Center at Lehigh Valley Hospital, Allentown, Pennsylvania
  - St. Luke's Hospital Cancer Center, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Easton Hospital, Easton, Pennsylvania
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - UPMC Cancer Center at Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - Mercy Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Williamsport Hospital, Williamsport, Pennsylvania
  - Women and Infants Hospital of Rhode Island, Providence, Rhode Island
  - Avera Sacred Heart Hospital, Yankton, South Dakota
  - Baptist Cancer Institute at Baptist Memorial Hospital - Memphis, Memphis, Tennessee
  - Sarah Cannon Cancer Center at Centennial Medical Center, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Vanderbilt Medical Center, Nashville, Tennessee
  - Baptist Hospital, Nashville, Tennessee
  - Seton Shivers Cancer Program at Brackenridge Hospital, Austin, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Zale Lipshy University Hospital, Dallas, Texas
  - Parkland Health and Hospital System, Dallas, Texas
  - St. Paul University Hospital, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas
  - Simmons Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Baylor University Medical Center - Houston, Houston, Texas
  - Doctor's Hospital of Laredo, Laredo, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Southwest Cancer and Research Center at University Medical Center, Lubbock, Texas
  - Cottonwood Hospital Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Dixie Regional Medical Center, St. George, Utah
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - Carilion New River Valley Medical Center, Christiansburg, Virginia
  - INOVA Fair Oaks Hospital, Fairfax, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Carilion Health System - Cancer Center of Western Virginia, Roanoke, Virginia
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - West Virginia University Hospitals, Morgantown, West Virginia
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Vince Lombardi Cancer Clinic at St. Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
- Peter MacCallum Cancer Centre, East Melbourne, Victoria, Australia
- CancerCare Manitoba, Winnipeg, Manitoba, Canada
- Ireland (2):
  - Cork University Hospital, Cork
  - St. Vincent's University Hospital, Dublin

REFERENCES:
- [Background] Ainsworth RK, Kollias J, Le Blanc A, De Silva P. The clinical impact of the American College of Surgeons Oncology Group Z-0011 trial--results from the BreastSurgANZ National Breast Cancer Audit. Breast. 2013 Oct;22(5):733-5. doi: 10.1016/j.breast.2012.11.005. Epub 2013 Jan 2. PMID 23290275
- [Background] Gainer SM, Hunt KK, Beitsch P, Caudle AS, Mittendorf EA, Lucci A. Changing behavior in clinical practice in response to the ACOSOG Z0011 trial: a survey of the American Society of Breast Surgeons. Ann Surg Oncol. 2012 Oct;19(10):3152-8. doi: 10.1245/s10434-012-2523-z. Epub 2012 Jul 21. PMID 22820938
- [Background] Olson JA Jr, McCall LM, Beitsch P, Whitworth PW, Reintgen DS, Blumencranz PW, Leitch AM, Saha S, Hunt KK, Giuliano AE; American College of Surgeons Oncology Group Trials Z0010 and Z0011. Impact of immediate versus delayed axillary node dissection on surgical outcomes in breast cancer patients with positive sentinel nodes: results from American College of Surgeons Oncology Group Trials Z0010 and Z0011. J Clin Oncol. 2008 Jul 20;26(21):3530-5. doi: 10.1200/JCO.2007.15.5630. PMID 18640934
- [Background] Leitch AM, McCall L, Beitsch P, et al.: Factors influencing accrual to ACOSOG Z0011, a randomized phase III trial of axillary dissection vs. observation for sentinel node positive breast cancer. [Abstract] J Clin Oncol 24 (Suppl 18): A-601, 2006.
- [Result] Krishnan MS, Recht A, Bellon JR, Punglia RS. Trade-offs associated with axillary lymph node dissection with breast irradiation versus breast irradiation alone in patients with a positive sentinel node in relation to the risk of non-sentinel node involvement: implications of ACOSOG Z0011. Breast Cancer Res Treat. 2013 Feb;138(1):205-13. doi: 10.1007/s10549-013-2418-0. Epub 2013 Jan 22. PMID 23338762
- [Result] Shah-Khan M, Boughey JC. Evolution of axillary nodal staging in breast cancer: clinical implications of the ACOSOG Z0011 trial. Cancer Control. 2012 Oct;19(4):267-76. doi: 10.1177/107327481201900403. PMID 23037494
- [Result] Caudle AS, Hunt KK, Kuerer HM, Meric-Bernstam F, Lucci A, Bedrosian I, Babiera GV, Hwang RF, Ross MI, Feig BW, Hoffman K, Litton JK, Sahin AA, Yang W, Hortobagyi GN, Buchholz TA, Mittendorf EA. Multidisciplinary considerations in the implementation of the findings from the American College of Surgeons Oncology Group (ACOSOG) Z0011 study: a practice-changing trial. Ann Surg Oncol. 2011 Sep;18(9):2407-12. doi: 10.1245/s10434-011-1593-7. No abstract available. PMID 21327455
- [Result] Giuliano AE, Hunt KK, Ballman KV, Beitsch PD, Whitworth PW, Blumencranz PW, Leitch AM, Saha S, McCall LM, Morrow M. Axillary dissection vs no axillary dissection in women with invasive breast cancer and sentinel node metastasis: a randomized clinical trial. JAMA. 2011 Feb 9;305(6):569-75. doi: 10.1001/jama.2011.90. PMID 21304082
- [Result] Giuliano AE, McCall L, Beitsch P, Whitworth PW, Blumencranz P, Leitch AM, Saha S, Hunt KK, Morrow M, Ballman K. Locoregional recurrence after sentinel lymph node dissection with or without axillary dissection in patients with sentinel lymph node metastases: the American College of Surgeons Oncology Group Z0011 randomized trial. Ann Surg. 2010 Sep;252(3):426-32; discussion 432-3. doi: 10.1097/SLA.0b013e3181f08f32. PMID 20739842
- [Result] Lucci A, McCall LM, Beitsch PD, Whitworth PW, Reintgen DS, Blumencranz PW, Leitch AM, Saha S, Hunt KK, Giuliano AE; American College of Surgeons Oncology Group. Surgical complications associated with sentinel lymph node dissection (SLND) plus axillary lymph node dissection compared with SLND alone in the American College of Surgeons Oncology Group Trial Z0011. J Clin Oncol. 2007 Aug 20;25(24):3657-63. doi: 10.1200/JCO.2006.07.4062. Epub 2007 May 7. PMID 17485711
- [Derived] Giuliano AE, Ballman KV, McCall L, Beitsch PD, Brennan MB, Kelemen PR, Ollila DW, Hansen NM, Whitworth PW, Blumencranz PW, Leitch AM, Saha S, Hunt KK, Morrow M. Effect of Axillary Dissection vs No Axillary Dissection on 10-Year Overall Survival Among Women With Invasive Breast Cancer and Sentinel Node Metastasis: The ACOSOG Z0011 (Alliance) Randomized Clinical Trial. JAMA. 2017 Sep 12;318(10):918-926. doi: 10.1001/jama.2017.11470. PMID 28898379
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/